CLINICAL TRIAL: NCT01354821
Title: Medical & Economical Evaluation of Endovascular Therapy of Complex Thoracal Abdominal Aneurysms (Type 1-3 Thoracal Abdominal Aneurysms) by Fenestrated & Branched Stent-grafts
Brief Title: Medical & Economical Evaluation of Fenestrated & Branched Stent-grafts to Treat Complex Thoracal Abdominal Aneurysms
Acronym: Windows2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P090209
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Aortic Aneurysm
Keywords: Aorta; Aneurysm; endovascular; stent-graft
MeSH Terms: conditions — Aortic Aneurysm; Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endovascular therapy branched (Active Comparator): Endovascular therapy branched or fenestrated stent-graft
  Interventions: Procedure: Endovascular aortic repair
- Open surgical repair (Other): Open surgical repair or aortic replacement with revascularization of visceral arteries
  Interventions: Procedure: Open surgical repair

INTERVENTIONS:
Procedure: Endovascular aortic repair — Insertion via bilateral femoral access, stent-graft deployment under fluoroscopic guidance, complementary stenting of visceral arteries, control angiogram
  Arms: Endovascular therapy branched
Procedure: Open surgical repair — Conventional therapy in France with the national database of the M.O.H.
  Arms: Open surgical repair

SUMMARY:
The aim of this study is to prospectively compare the perioperative mortality severe morbidity and the costs of endovascular versus conventional surgical repair of type 1, 2 and 3 thoracal abdominal aortic aneurysms.

DETAILED DESCRIPTION:
The aim of this study is to prospectively compare the perioperative mortality severe morbidity and the costs of endovascular versus conventional surgical repair of type 1, 2 and 3 thoracal abdominal aortic aneurysms.

The primary goal of the study is to demonstrate a significant drop in 30-day mortality and life threatening morbidity in the endovascular arm of the study. Our hypothesis, derived from the literature, that the average 30-days mortality is 3% after endovascular repair and 10% after open surgery justifies the design of a prospective study between endovascular therapy (50 patients (amendment n.5 - 9/07/2013) treated in 5 University hospitals with significant experience of the technique) and open repair (220 similar patients analyzed from the national database of the MOH).

In-hospital morbidity are similarly expected to be lower in the endovascular group. The investigators also wish to demonstrate that endovascular repair does not represent a significant overcost, as compared to open repair. The cost of the implantable medical device (IMD), of follow-up screening, and of eventual repeated interventions should be compensated by a reduced stay in intensive care unit ICU, and by a reduced in-hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

The following anatomical inclusion criteria must be met:

* Absence of significant angulations (< 60°) of aorta or of iliac arteries
* Absence of tight stenosis (>70%) of more than one target artery (renal or visceral artery to be perfused from the side holes of the stent-graft)
* Diameter of target arteries over 5 mm
* Iliac and femoral arteries allowing insertion of the delivery system (> 7 mm) or suitable for insertion of an access conduit

Exclusion Criteria:

* Limited expected life expectancy
* Emergency cases
* Refuse to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-11; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 30-day postoperative

SECONDARY OUTCOMES:
complications | 30-day postoperative
Length of Intensive Care Unit (ICU) stay | 30-day postoperative
Length of Hospital stay | 30-day postoperative
Overall cost | 30-day postoperative
Reinterventions | 2-year follow up
Global survival | 2-year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Becquemin, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Amiot S, Haulon S, Becquemin JP, Magnan PE, Lermusiaux P, Goueffic Y, Jean-Baptiste E, Cochennec F, Favre JP; Association Universitaire de Recherche en Chirurgie Vasculaire. Fenestrated endovascular grafting: the French multicentre experience. Eur J Vasc Endovasc Surg. 2010 May;39(5):537-44. doi: 10.1016/j.ejvs.2009.12.008. Epub 2010 Jan 25. PMID 20093051